CLINICAL TRIAL: NCT01213433
Title: Amodiaquine+Artesunate for the Treatment of Uncomplicated Falciparum Malaria in Nanoro, Burkina Faso
Brief Title: Amodiaquine+Artesunate for Uncomplicated Malaria Treatment
Acronym: ASAQ-MAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Muraz (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Tinto Halidou, PharmD, PhD, Centre Muraz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 016-2010
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Uncomplicated Malaria
MeSH Terms: interventions — amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amodiaquine+Artesunate (Experimental)
  Interventions: Drug: Artesunate-Amodiaquine

INTERVENTIONS:
Drug: Artesunate-Amodiaquine — Coformulated AQ+AS by Sanofi-Aventis has been pre-qualified by WHO in 2008.It is administered once daily for three consecutive days, and it is available in three different dosages (25mg/67.5mg; 50mg/135mg; 100mg/270mg)

SUMMARY:
This is a phase IV one-arm study aiming at recruiting 50 patients to assess the efficacy of AQ+AS in patients with a positive RDT diagnosis of malaria in Nanoro, Burkina Faso.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged 6 months and above.
* Body weight of 5 Kg and above.
* RDT positive test.
* Fever (axillary temperature at ≥ 37.5°C) or history of fever in the previous 24 hours.
* Signed (or thumb-printed whenever patients are illiterate) informed consent.
* Patients' willingness and ability to comply with the study protocol for the duration of the study.

Exclusion Criteria:

* Participation in any other investigational drug study (antimalarial or others) during the previous 30 days.
* Known hypersensitivity to the study drugs.
* Severe malaria.
* Danger signs: not able to drink or breast-feed, vomiting (> twice in 24hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand.
* Known intercurrent illness or any condition (cardiac, renal, hepatic diseases) which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.
* Severe malnutrition (defined as weight for height <70% of the median NCHS/WHO reference).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Treatment failure at day 28 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRUN, Nanoro, Boulkiemdé, Burkina Faso